CLINICAL TRIAL: NCT01267357
Title: Expression of the P16 Protein in Serous Papillary Endometrial Cancer, and Its Clinical and Prognostic Significance
Brief Title: P16 Staining as Prognostic Biomarker in Serous Papillary Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr. Itamar Netzer, Rambam Medical Center
Other Study IDs: 230CTIL
Record Dates: First submitted 2010-12-15; First posted 2010-12-28 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-11

CONDITIONS: Serous Papillary Endometrial Cancer
Keywords: Serous Papillary Endometrial Cancer; Endometrioid endometrial cancer; biomarkers; P16; P53; Prognosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Existing paraffin pathology blocks in hospital's library were used. Remainder of material was returned to the library.
  No identifying features were retained or attached to specimens.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Serous papillary endometrial ca patients: 30 patients diagnosed with SP endometrial ca
  Interventions: Other: no intervention
- Endometrioid endometrial ca: 32 patients diagnosed with Endometrioid endometrial ca
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
P16 is a tumor suppressor protein implicated in serous papillary endometrial carcinoma. Evidence from previous trials indicates that it may be used as a diagnostic biomarker distinguishing this disease from endometrioid endometrial cancer. Additional evidence points to its prognostic value.

The current study will evaluate p16 both as a diagnostic tool for serous papillary endometrial cancer and as a prognostic biomarker.

following anonymization, histology blocks will be microtomed and stained for P16 and P53 proteins.

Blocks from endometrioid endometrial cancer will be used as a control group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of endometrial cancer
* histology block exists in hospital's library

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women diagnosed with endometrial cancer, having undergone surgery and having received chemotherapy in our institution.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | last followup (2-10 years)

SECONDARY OUTCOMES:
progression free survival | Current follow up (2-10 years)
correlation of P16 stain with histological diagnosis | at last follow up (2-10 years)

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel